CLINICAL TRIAL: NCT06060717
Title: Evaluation of the F&P Caramel Nasal Mask, US, 2023
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Fisher and Paykel Healthcare (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CIA-337
Record Dates: First submitted 2023-09-24; First posted 2023-09-29 (Actual); Results first posted 2025-09-23 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-09

CONDITIONS: Obstructive Sleep Apnea
MeSH Terms: conditions — Sleep Apnea, Obstructive

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: No

ARMS (1):
- Single-arm, non-randomised open-label (Other)
  Interventions: Device: F&P Caramel

INTERVENTIONS:
Device: F&P Caramel — Nasal mask

SUMMARY:
The purpose of this clinical investigation is to evaluate the performance and safety of the F&P Caramel nasal mask in a home environment.

ELIGIBILITY:
Inclusion Criteria:

* Persons who are ≥22 years of age
* Persons who weigh ≥66 pounds
* Persons who have been prescribed PAP therapy by a physician
* Persons who are existing nasal mask or sub-nasal mask users with ≥3 months of use prior to enrolment in the clinical trial
* Persons who are compliant with PAP therapy for ≥4 hours per night for ≥70% of nights for a 14-day period within 30 days prior to enrolment in the clinical trial
* Persons who are fluent in spoken and written English
* Persons who possess the capacity to provide informed consent

Exclusion Criteria:

* Persons who are intolerant to PAP therapy
* Persons who possess, or suffer from, anatomical or physiological conditions which make PAP therapy inappropriate
* Persons who are required to use PAP therapy for >12 hours per day or for extensive periods, not including sleep or naps
* Persons who are trying to get pregnant, are pregnant, or think they may be pregnant
* Persons who have an IPAP pressure of >30 cmH2O if on BPAP
* Persons who use a PAP therapy device for the delivery of medicines, except supplemental oxygen
* Persons who use a PAP therapy device that does not possess data recording capabilities to capture AHI and a numerical indicator of leak that is accessible to the investigation site

Min Age: 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 45 (Actual)
Dates: Start 2023-11-27 (Actual); Primary Completion 2023-12-11 (Actual); Study Completion 2024-06-11 (Actual)

CONTACTS AND LOCATIONS:
Locations (1):
- Clayton Sleep Institute, St Louis, Missouri, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Caramel Nasal Mask: Participants to use nasal mask for 14 days. Caramel Nasal Mask:Nasl mask for the treatment of obstructive sleep apnea (OSA)
Period: Overall Study
Arm/Group | Caramel Nasal Mask
Started | 45
Completed | 43
Not Completed | 2

BASELINE CHARACTERISTICS:
Population: Participants with obstructive sleep apnea (OSA) that have been been prescribed positive airway pressure (PAP) therapy
Groups:
- F&P Caramel: Nasal Mask: Participants to use nasal mask for 14 days. Caramel Nasal Mask: Nasal mask for the treatment of obstructive sleep apnea (OSA).
Arm/Group | F&P Caramel: Nasal Mask
Number analyzed (Participants) | 43
Age, Customized [Count of Participants; unit: Participants] | 43
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 18
  Male | 25
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 4
  Not Hispanic or Latino | 39
  Unknown or Not Reported | 0

OUTCOME MEASURES:

1. Primary Outcome: Therapeutic Efficacy
Description: Determined by Apnea-Hypopnea Index (AHI) recorded on PAP therapy machines after 14 days of use. The Apnea-Hypopnea index (AHI) is the sum of the apneas and hypopneas divided by the hours of sleep. AHI values are typically categorized as 5-15/hr = mild; 15-30/hr = moderate; and >= 30/h = severe AHI is measured by dividing the total number of recorded apneas (complete breathing stops) and hypopneas (shallow breathing episodes) by the total number of hours a person slept during an overnight sleep study or using a PAP device.
  Higher AHI values represent worse outcomes. There is no maximum theoretical index score.
Time Frame: Baseline and14±5 days
Measure: Mean (Full Range); unit: events per hour
Groups:
- F&P Caramel: Nasal Mask: Determined by Apnea-Hypopnea Index (AHI) recorded on PAP therapy machines after 14 days of use.
Arm/Group | F&P Caramel: Nasal Mask
Number analyzed (Participants) | 43
events per hour | 1.69 [0.2 to 17.3]

2. Primary Outcome: Epworth Sleepiness Scale
Description: All relevant time points used in the calculation in the Time Frame (e.g., baseline and 14±5 days).
  Note: change was calculated from two time points as the value at the later time point minus the value at the earlier time point (e.g., value at 14±5 days minus value at baseline).
  Change between two time points is reported. Scale range: 0 (minimum score) to 24 (maximum score) (higher scores represent worse outcomes)
Time Frame: Baseline and14±5 days
Measure: Mean (Full Range); unit: Epworth Sleepiness Score (ESS)
Groups:
- F&P Caramel: Nasal Mask: Participants to use nasal mask for 14 days. Caramel Nasal Mask:Nasal mask for the treatment of obstructive sleep apnea (OSA)
Arm/Group | F&P Caramel: Nasal Mask
Number analyzed (Participants) | 43
Epworth Sleepiness Score (ESS) | 7 [0 to 13]

ADVERSE EVENTS:
Time Frame: 14 days
Arm/Group | F&P Caramel: Nasal Mask
All-Cause Mortality (participants affected / at risk) | 0/43
Serious Adverse Events (participants affected / at risk) | 0/43
Other Adverse Events (participants affected / at risk) | 4/43
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | F&P Caramel: Nasal Mask (N=43)
Common Cold (Respiratory, thoracic and mediastinal disorders) | 4 (4)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2023-10-18): https://cdn.clinicaltrials.gov/large-docs/17/NCT06060717/Prot_SAP_000.pdf